CLINICAL TRIAL: NCT00519233
Title: A Phase I Investigation of the Intravenous Administration of AGS-1C4D4 in Patients With Advanced Hormone Refractory Prostate Cancer
Brief Title: AGS-1C4D4 in Patients With Advanced Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Agensys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007001; MK4721-003; 2007_535
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Prostate Cancer
Keywords: HRPC; Advanced hormone refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — MK-4721

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1.AGS-1C4D4 (Experimental)
  Interventions: Drug: AGS-1C4D4

INTERVENTIONS:
Drug: AGS-1C4D4 — IV

SUMMARY:
The present study will investigate the safety, tolerability and spectrum of side effects of AGS-1C4D4. As such, this study will characterize the dose limiting toxicities (DLT) and potentially the maximum tolerated dose (MTD) of AGS-1C4D4 in patients with advanced HRPC.

DETAILED DESCRIPTION:
Cohorts of 1-6 patients will be administered AGS-1C404 in sequentially rising dose levels. Dose escalation will continue until the MTD of AGS-1C4D4 is established or the maximum planned dose is reached.

ELIGIBILITY:
Inclusion Criteria:

* Patient has hormone-refractory metastatic prostate cancer

Exclusion Criteria:

* Patient has had chemotherapy, radiotherapy, or biological therapy within the past 4 weeks or has not recovered from side effects
* Patient is currently participating or has participated in an investigational study within the past 30 days
* Patient has illness or circumstance that could limit compliance with the study requirements
* Patient uses illicit drugs or had a recent history of drug or alcohol abuse within the last year
* Patient has Hepatitis B or C

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability and side effects of AGS-1C4D4 in adult patients with advanced HRPC. | 3 Months

SECONDARY OUTCOMES:
The pharmacokinetic profile of AGS-1C4D4 in adult patients with advanced HRPC. | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Agensys, Inc.
Locations (2):
- United States (2):
  - Baltimore, Maryland
  - New York, New York

REFERENCES:
- [Background] Antonarakis ES, Carducci MA, Eisenberger MA, Denmeade SR, Slovin SF, Jelaca-Maxwell K, Vincent ME, Scher HI, Morris MJ. Phase I rapid dose-escalation study of AGS-1C4D4, a human anti-PSCA (prostate stem cell antigen) monoclonal antibody, in patients with castration-resistant prostate cancer: a PCCTC trial. Cancer Chemother Pharmacol. 2012 Mar;69(3):763-71. doi: 10.1007/s00280-011-1759-9. Epub 2011 Oct 22. PMID 22020316